CLINICAL TRIAL: NCT06400719
Title: An Open Label, Single Arm Pilot Study to Investigate the Safety and Tolerability of a Single 300mg Intravenous Dose of AVT16 in Healthy Adult Subjects Aged 18 to 55 Years Inclusive
Brief Title: Pilot Study of AVT16 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVT16-GL-F01
Record Dates: First submitted 2024-04-24; First posted 2024-05-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AVT16 (Experimental): Single intravenous administration of 300mg AVT16, proposed biosimilar to vedolizumab
  Interventions: Biological: AVT16

INTERVENTIONS:
Biological: AVT16 — Single intravenous administration of 300mg of AVT16

SUMMARY:
This is a pilot study in healthy adult subjects to evaluate the safety and tolerability of AVT16 after administration of a single intravenous administration. Pharmacokinetics and immunogenicity of AVT16 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged between 18 and 55 years old inclusive
* Medical history without evidence of clinically significant disorder, condition or disease that would pose a risk to subject safety
* Haematology and biochemistry tests within normal range

Exclusion Criteria:

* History of relevant drug and/or food allergies
* History of hypersensitivity to vedolizumab, AVT16 of their constituents
* Past or concurrent medical conditions that could potentially increase subject's risks or interfere with study evaluations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Incidence, nature and severity of Treatment Emergent Adverse Events | 18 weeks
  Safety and Tolerability of AVT16

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of AVT16 | 18 weeks
  Pharmacokinetic parameters
Frequency of anti-drug antibodies | 18 weeks
  Immunogenicity of AVT16

CONTACTS AND LOCATIONS:
Locations (1):
- CCST, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No